CLINICAL TRIAL: NCT02370394
Title: Computer-Based Intervention for Victimized Perinatal Women With Mental Illness (Phase 1)
Brief Title: Intervention for IPV Perinatal Women- RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Director of Behavioral Medicine Research, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0056; 1R21HD077358-01A1 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Intimate Partner Violence
Keywords: Intimate Partner Violence; Perinatal Women; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROSE Program (Experimental): Participants received a 35-40-minute intervention on the Tablet PC and an in-person 10-15-minute booster session conducted by interventionists within a month after the intervention. Participants in this condition completed a baseline assessment as well as a follow-up assessment 3 months later.
  Interventions: Behavioral: ROSE Program
- Control Condition (No Intervention): Control Condition consisted of a series of questions regarding television show preferences and then viewed a brief series of videos of popular entertainers/shows, with subsequent requests for ratings of subjective preference. Participants in this condition completed a baseline assessment as well as a follow-up assessment 3 months later.

INTERVENTIONS:
Behavioral: ROSE Program — The ROSE Program was specifically tailored, innovative and relevant to diverse, racial and ethnic perinatal women in a number of ways including the images and content used in the intervention and coordinating study appointments with treatment visits. It was tailored to the current IPV risk assessment, pregnancy or postpartum status of each participant, was designed to reach participants across levels of motivation for change. The content of ROSE was theory-driven, consistent with the Motivational Interviewing model of behavior, and consistent with the literature on effective interventions that address IPV.
  Arms: ROSE Program

SUMMARY:
The study developed and assessed an innovative, high-reach, easily implementable, low-cost computer-delivered intervention (Reach out for a Safe Environment; ROSE Program) that addressed known barriers in early identification and intervention with perinatal women with IPV seeking treatment for mental illness.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a significant social and public health problem among perinatal women. Research suggests that from 21% to 33% of perinatal women report IPV and there is an enormous amount of morbidity associated with IPV. Moreover, IPV places a woman at high risk for several psychiatric disorders, which transforms the perinatal period from an already challenging process into a potentially overwhelming one. Further, IPV and untreated mental illness during the perinatal period pose a dual risk of adverse physical and emotional outcomes for women and their developing fetus/infant. Experts in the field advocate for more IPV screening and intervention to take place among women who are at high-risk for IPV. Given the high rates of IPV among women who seek mental health treatment, mental health clinics compared to other medical settings (e.g. primary care) are more effective sites for focused case finding and intervention. Further, the presence of IPV increases the likelihood of disengagement from treatment, which could compromise the ability of women with IPV to effectively use important shelter and community resources necessary for establishing safety for themselves and their children. A timely intervention might reduce the risk of future IPV, improve treatment utilization, and reduce mental health symptoms. A brief intervention that is designed specifically for the unique needs of perinatal women with IPV seeking mental health treatment provides a tremendous opportunity to intervene with a group of women who are particularly vulnerable and who might be unusually open to making changes to their lives.

This study is the first step towards developing a computer-based brief intervention ("Reach Out for a Safe Environment") that targets intimate partner violence in perinatal women in mental health treatment and constitutes the developmental aims of a larger study. The aims were to perform a small open trial (n = 8) of the Reach Out for a Safe Environment (ROSE) intervention to assess feasibility of recruitment of target population and acceptability of intervention and study procedures. Also, to conduct a randomized controlled pilot study in a sample of 50 perinatal women seeking mental health treatment who screen positive for recent IPV to demonstrate the acceptability and feasibility of the ROSE intervention via participant report of ease of use, helpfulness, and overall satisfaction.

We collected several measures on the feasibility of the research design, the acceptability of ROSE, and on intervention effects for IPV severity and level of self-care strategies (primary outcomes), motivation and self efficacy (secondary outcomes), and use of recommended mental health treatment services (tertiary outcome). This phase used a two-group, randomized, controlled design with an initial session for both conditions plus booster session one month later for the intervention condition. The initial intervention session was conducted close to an intake visit for mental health difficulties, with a booster session within one month following baseline. There was a 3-month follow up assessment. Assessments and the booster session were conducted in a private room or at a location that was a convenient location for the woman and one that provided a confidential, safe, and comfortable environment for the participant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or postpartum women (up to 6 months after delivery)
* Age 18 or older
* Seeking mental health treatment at The Center for Women's Behavioral Health (WBH) at Women and Infants Hospital (WIH)
* Endorsed any IPV during the past 12 months as measured by the Woman Abuse Screening Tool (WAST)

Exclusion Criteria:

* Inability to provide informed consent (e.g., due to psychosis, intoxication, or other clear cognitive impairment)
* Inability to understand English (understand the consent form when read aloud and assessments that are narrated by computer)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Women and Infants' Hospital
Locations (1):
- Center for Women's Behavioral Health at Women and Infants' Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Zlotnick C, Tzilos Wernette G, Raker CA. A randomized controlled trial of a computer-based brief intervention for victimized perinatal women seeking mental health treatment. Arch Womens Ment Health. 2019 Jun;22(3):315-325. doi: 10.1007/s00737-018-0895-1. Epub 2018 Aug 7. PMID 30088145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited perinatal women from The Center for Women's Behavioral Health (WBH) at Women and Infants Hospital (WIH) between May 2015 and April 2016.
Groups:
- ROSE Program: Participants received a 50-minute intervention on the Tablet PC immediately after their baseline assessment and an in-person 30-minute booster session conducted by interventionists within a month after the intervention. There was also a follow-up assessment 3 months after completion of the ROSE program.
  ROSE Program: The ROSE Program was specifically tailored, innovative and relevant to diverse, racial and ethnic perinatal women in a number of ways including the images and content used in the intervention and coordinating study appointments with treatment visits. It was also tailored on the current IPV risk assessment, pregnancy or postpartum status of each participant, was designed to reach participants across levels of motivation for change. The content of ROSE was theory-driven, consistent with the Motivational Interviewing model of behavior, and consistent with the literature on effective interventions that address IPV.
- Control Condition: Control Condition consisted of a series of questions regarding television show preferences and viewing a brief series of videos of popular entertainers/shows, with subsequent requests for ratings of subjective preference. Participants in this condition completed a baseline assessment as well as a follow-up assessment 3 months later.
Period: Overall Study
Arm/Group | ROSE Program | Control Condition
Started | 28 | 25
Completed | 26 | 23
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ROSE Program | Control Condition | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 27 | 24 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.03 [18 to 37] | 28.32 [18 to 36] | 27.64 [18 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite Abuse Scale (CAS)-CAS Victimization Total Score
Description: A widely used self-report of behaviors that includes a 36-item scale - only the CAS Victimization Total score was calculated. Items were scored between 0 and 5, with Never=0 and Daily=5. Scale range is from 0-180. Mean score was used to calculate differences between baseline and follow-up and between groups. The lower the score, the better or less victimization.
Time Frame: Assessed at baseline, and again three months later
Population: The number of participants analyzed differs from baseline to follow-up because 2 dropped out of the ROSE intervention group, and 1 dropped out and 1 withdrew (no longer interested) from the control condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROSE Program | Control Condition
Number analyzed (Participants) | 28 | 25
units on a scale
  CAS at Baseline | 26.36 (17.81) | 16.56 (12.25)
  CAS at Follow-up: number analyzed (Participants) | 26 | 23
  CAS at Follow-up | 12.38 (12.44) | 16.52 (20.23)
Statistical Analysis 1: Comparison: ROSE Program vs Control Condition; CAS Victimization Total Score at Follow Up; Test type: Superiority; p = 0.4016, t-test, 2 sided; Unequal variances handled by Satterthwaite's degrees of freedom; Mean Difference (Final Values) = -4.14, 95% CI 2-sided [-14.02 to 5.75]
Statistical Analysis 2: Comparison: ROSE Program vs Control Condition; Change in CAS Victimization Total score from Baseline to Follow Up; Test type: Superiority; p = 0.0072, t-test, 2 sided; Mean Difference (Net) = 14.46, 95% CI 2-sided [4.11 to 24.82]

2. Primary Outcome: Safety Behavior Checklist (SBC)
Description: Includes 15 items that assess the use of strategies suggested to keep victim safe (e.g., hiding money and extra clothing). Items were scored as Yes=1 or No=0 or Not applicable. Scale range is from 0-15. Mean score was used to calculate differences between baseline and follow-up and between groups. The higher the score, the better or more use of safety behaviors.
Time Frame: Assessed at baseline, and again three months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROSE Program | Control Condition
Number analyzed (Participants) | 28 | 25
units on a scale
  SBC at Baseline | .28 (.23) | .36 (.23)
  SBC at Follow Up: number analyzed (Participants) | 26 | 23
  SBC at Follow Up | .28 (.28) | .32 (.29)
Statistical Analysis 1: Comparison: ROSE Program vs Control Condition; Safety Behavior Change Score at Follow Up; Test type: Superiority; p = 0.6011, t-test, 2 sided; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.21 to 0.12]
Statistical Analysis 2: Comparison: ROSE Program vs Control Condition; Change is Safety Behavior Change Score from Baseline to Follow Up; Test type: Superiority; p = 0.9116, t-test, 2 sided; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.16 to 0.15]

3. Primary Outcome: Effectiveness in Obtaining Resources Scale (EOR)
Description: Assesses the women's effectiveness in obtaining resources from 11 different types of community resources including mental health treatment, church or clergy, health care, legal services, police, or social services. Items were scored as Yes=1 or No=0. Scale range is from 0-11. Mean score was used to calculate differences between baseline and follow-up and between groups. The higher the score, the better or more they were effective in obtaining resources.
Time Frame: Assessed at baseline, and again three months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROSE Program | Control Condition
Number analyzed (Participants) | 28 | 25
units on a scale
  EOR at Baseline | 2.46 (1.71) | 3.48 (2.87)
  EOR at Follow Up: number analyzed (Participants) | 26 | 23
  EOR at Follow Up | 3.31 (2.59) | 3.43 (2.59)
Statistical Analysis 1: Comparison: ROSE Program vs Control Condition; EOR Number of issues Effective at Accomplishing at Follow Up; Test type: Superiority; p = 0.8646, t-test, 2 sided; Unequal variances handled by Satterthwaite's degrees of freedom; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-1.62 to 1.36]
Statistical Analysis 2: Comparison: ROSE Program vs Control Condition; Change in Number of Issues Effective at Accomplishing from Baseline to Follow Up; Test type: Superiority; p = 0.3045, t-test, 2 sided; Mean Difference (Net) = -0.86, 95% CI 2-sided [-2.54 to 0.82]

4. Secondary Outcome: Motivation Scale
Description: A 1-item measure, was modified to assess how ready they are to use treatment, resources, and/or support for any partner abuse. This item was scored with a range from 0-10. 0=not ready at all to 10=completely ready. Mean score was used to calculate differences between baseline and follow-up and between groups. The higher the score, the better or more ready to use treatment, resources, or support for any partner abuse.
Time Frame: Assessed at baseline, and again three months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROSE Program | Control Condition
Number analyzed (Participants) | 28 | 25
units on a scale
  Motivation Scale at Baseline | 6.18 (2.76) | 7.52 (3.48)
  Motivation Scale at Follow Up: number analyzed (Participants) | 26 | 23
  Motivation Scale at Follow Up | 6.81 (3.64) | 7.22 (3.15)
Statistical Analysis 1: Comparison: ROSE Program vs Control Condition; Motivation Scale at Follow Up; Test type: Superiority; p = 0.9085, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ROSE Program vs Control Condition; Change in Motivation Scale from Baseline to Follow Up; Test type: Superiority; p = 0.3256, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: The Readiness to Change Contemplation Ladder
Description: One item measure to assess readiness to make changes to increase safety. This item was scored with a range from 0-10. 0=not prepared to change to 10=already changing. Mean score was used to calculate differences between baseline and follow-up and between groups. The higher the score, the better or more ready to make changes to increase safety.
Time Frame: Assessed at baseline, and again three months later
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ROSE Program | Control Condition
Number analyzed (Participants) | 28 | 25
units on a scale
  Readiness at Baseline | 8.25 (2.01) | 8.08 (2.68)
  Readiness at Follow Up: number analyzed (Participants) | 26 | 23
  Readiness at Follow Up | 8.00 (2.94) | 7.26 (2.97)
Statistical Analysis 1: Comparison: ROSE Program vs Control Condition; Readiness at Follow Up; Test type: Superiority; p = 0.4085, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ROSE Program vs Control Condition; Change in Readiness from Baseline to Follow Up; Test type: Superiority; p = 0.2467, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between the date of the baseline and the 3 month follow-up, generally for 3 months, depending on when the participant's 3 month follow-up actually occurred.
Description: The DSMB decided that the following would be included as SAEs: any serious/life threatening threats of intimate partner violence, rape, sexual assault, emergency room visits as well as death, hospitalization, and life-threatening events, as described in the clinicaltrials.gov definitions.
Arm/Group | ROSE Program | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 9/28 | 6/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ROSE Program (N=28) | Control Condition (N=25)
Hospitalization-general medical issue (Surgical and medical procedures) | 4 (4) | 2 (2)
Hospitalization-inpatient-psyc (Psychiatric disorders) | 3 (3) | 1 (1)
IPV-no medical care (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) — Physical abuse or rape - no medical care sought for injuries
IPV related emergency room visit (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes